CLINICAL TRIAL: NCT07172555
Title: The Role Of Virtual Dietetic Interventions In Patients With Coeliac Disease
Brief Title: Virtual Dietetic Interventions in Patients With Coeliac
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH22680
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Coeliac Disease
Keywords: coeliac disease; diet; webinar
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Dietetic First-Appointment Webinar for Coeliac Disease (Experimental): Participants allocated to this arm will receive a pre-recorded, dietitian-led "first appointment" webinar designed specifically for adults newly diagnosed with coeliac disease. The webinar will provide comprehensive education on the gluten-free diet, approaches to avoid cross-contamination, and strategies for nutritional adequacy. The intervention allows participants to watch and re-watch the webinar at their convenience. All participants will undergo baseline assessments and will complete knowledge and satisfaction questionnaires immediately post-intervention, with follow-up clinical and patient-reported outcomes collected at 6 months.
  Interventions: Other: Virtual Dietetic First-Appointment Webinar for Coeliac Disease
- Standard Dietetic Consultation (Face-to-Face or Telephone) (Active Comparator): Participants in this group are allocated to receive the existing standard of care: an individual appointment with a specialist dietitian, delivered either in person (face-to-face) or by telephone. During the appointment, the dietitian provides a comprehensive overview of the gluten-free diet, strategies for avoiding cross-contamination, and advice on nutritional adequacy. As in the experimental arm, baseline assessment and validated questionnaires are administered pre- and post-intervention, with follow-up at 6 months to collect clinical, adherence, satisfaction, and quality of life data for direct comparison with the on-demand webinar intervention.
  Interventions: Other: Standard Dietetic Consultation (Face-to-Face or Telephone)

INTERVENTIONS:
Other: Virtual Dietetic First-Appointment Webinar for Coeliac Disease — This intervention is a dietitian-led, pre-recorded on-demand webinar specifically designed for adults who have been newly diagnosed with coeliac disease. It acts as a patient's first formal dietetic appointment after diagnosis and provides comprehensive education about coeliac disease and the strict gluten-free diet required for its management. Unlike traditional approaches, which rely on face-to-face or telephone appointments with a dietitian-and which often involve significant waiting times-the webinar is available immediately online, allowing patients to access trusted, specialist information at their own pace and convenience, including the opportunity to re-watch as needed
  Arms: Virtual Dietetic First-Appointment Webinar for Coeliac Disease
Other: Standard Dietetic Consultation (Face-to-Face or Telephone) — Participants in this group are allocated to receive the existing standard of care: an individual appointment with a specialist dietitian, delivered either in person (face-to-face) or by telephone. During the appointment, the dietitian provides a comprehensive overview of the gluten-free diet, strategies for avoiding cross-contamination, and advice on nutritional adequacy. As in the experimental arm, baseline assessment and validated questionnaires are administered pre- and post-intervention, with follow-up at 6 months to collect clinical, adherence, satisfaction, and quality of life data for direct comparison with the on-demand webinar intervention.
  Arms: Standard Dietetic Consultation (Face-to-Face or Telephone)

SUMMARY:
This clinical study is exploring whether a pre-recorded, on-demand webinar led by specialist dietitians can be as effective as traditional one-on-one appointments in helping people newly diagnosed with coeliac disease learn to follow a gluten-free diet. Coeliac disease is a serious, life-long condition where eating even tiny amounts of gluten, a substance found in wheat, barley, and rye, can cause damaging symptoms and long-term health problems. The only current treatment is sticking to a strict gluten-free diet, which can be difficult without proper support and guidance from dietitians.

The number of people being diagnosed with coeliac disease in the UK is growing, and this is placing extra pressure on NHS dietetic services, which are already stretched. Many patients currently face long waits or do not get any dietetic support at all. To address this, the research team at Sheffield Teaching Hospitals has developed an on-demand, first-appointment webinar to provide immediate access to trusted dietary information, with the aim of improving patient care and saving NHS resources.

In this study, adults newly diagnosed with coeliac disease at Sheffield Teaching Hospitals will be asked to join one of two groups: one group will receive their first dietitian appointment through the new on-demand webinar, while the other group will have a traditional face-to-face or phone appointment with a dietitian. Both groups will complete short questionnaires to measure their knowledge about the gluten-free diet, their symptoms, how well they are following the diet, and their quality of life, both before and after receiving their dietary support, and again after six months. Blood tests will also be used to monitor health markers.

The main goal of the research is to find out if the first-appointment webinar is just as effective as traditional appointments in helping patients understand and follow a gluten-free diet, feel satisfied with the support they receive, and achieve good health outcomes. If the study shows that the webinar approach is as good as traditional care, it could mean quicker, easier, and more consistent access to essential dietary support for people with coeliac disease, both locally and across the UK.

Hypothesis:

The study hypothesis is that a dietitian-led, on-demand, pre-recorded webinar for a first appointment is as effective as traditional one-to-one consultations (face-to-face or by phone) in helping newly diagnosed coeliac patients achieve the same standard health outcomes, dietary knowledge, and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years and over with serology- or biopsy-proven coeliac disease.

Exclusion Criteria:

Patients under the age of 18 years. Patients unable to provide written informed consent. Patients who are unable to understand or speak English. Patients unable to access digital resources. Poly-diagnosis that requires additional nutritional intervention (i.e. Diabetes or Inflammatory Bowel Disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge of Gluten-Free Diet | Baseline (pre-intervention), immediately post-intervention, and at 6-month follow-up.
  Assessed using the Coeliac Disease and Gluten-Free Diet Quiz, a structured and previously validated questionnaire administered at baseline, immediately post-intervention, and at 6 months. This tool evaluates patient knowledge related to coeliac disease and the gluten-free diet requirements for effective disease management. Scores pre- and post-intervention (webinar or standard care) will be compared to determine the educational impact of each modality.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie published results will be made available to researchers upon reasonable request following completion of the trial and publication of the main findings. Data will be stored securely and released only with appropriate approvals, in accordance with the Data Protection Act 2018 and Sheffield Teaching Hospitals NHS Trust policies. Requests for access may come from both internal and external research collaborators, and all IPD will be stripped of direct patient identifiers prior to sharing.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Rej A, Trott N, Kurien M, Branchi F, Richman E, Subramanian S, Sanders DS. Is Peer Support in Group Clinics as Effective as Traditional Individual Appointments? The First Study in Patients With Celiac Disease. Clin Transl Gastroenterol. 2020 Jan;11(1):e00121. doi: 10.14309/ctg.0000000000000121. PMID 31977451
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Rej A, Buckle RL, Shaw CC, Trott N, Urwin H, McGough N, Aziz I, Sanders DS. National survey evaluating the provision of gastroenterology dietetic services in England. Frontline Gastroenterol. 2020 Jun 16;12(5):380-384. doi: 10.1136/flgastro-2020-101493. eCollection 2021. PMID 35401953
- [Background] Caio G, Volta U, Sapone A, Leffler DA, De Giorgio R, Catassi C, Fasano A. Celiac disease: a comprehensive current review. BMC Med. 2019 Jul 23;17(1):142. doi: 10.1186/s12916-019-1380-z. PMID 31331324

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT07172555/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT07172555/ICF_001.pdf